CLINICAL TRIAL: NCT06246708
Title: Cultural Adaptation of a Self-help App for Grieving Syrian Refugees in Switzerland. A Feasibility and Acceptability Pilot-RCT
Brief Title: Cultural Adaptation of a Self-help App for Grieving Syrian Refugees in Switzerland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Transfusion SRC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBISYR
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Bereavement
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Pilot RCT with an intervention group and a wait-list control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive intervention at baseline for 5 weeks
  Interventions: Other: Self-help app with information for grieving Syrian Refugees
- Wait-list Control Group (Other): Participants receive the intervention after 5 weeks
  Interventions: Other: Wait-list

INTERVENTIONS:
Other: Self-help app with information for grieving Syrian Refugees — This study explores a self-help app for grieving Syrian refugees in Switzerland, featuring five chapters on grief, resources, space, negative thoughts, and future self-help. The Arabic app includes psychoeducational content, audio exercises, and videos. Users personalize it, save favorites, and set reminders. Tailored for Arabic-speaking refugees, it's accessible on iOS and Android, without invasive components. Participants complete one weekly chapter over five weeks. Data input is stored without manipulation. Accessible data includes completed chapters, subchapters, and feedback. The app promotes self-help, respecting cultural nuances for user engagement.
  Arms: Intervention Group
Other: Wait-list — Participants in the wait-list control group, receive access to the same intervention described above after a waiting period of 5 weeks.
  Arms: Wait-list Control Group

SUMMARY:
The goal of this pilot RCT is to investigate the acceptability and feasibility of an unguided culturally adapted self-help app for grieving Syrian refugees in Switzerland. Furthermore, the study will examine whether using the app has an effect on secondary outcomes (e.g., grief symptoms).The main questions it aims to answer are:

* Is the self-help app culturally acceptable and feasible in this target group and what do we need to adapt?
* Does the use of the self-help app reduce grief symptoms? (amongst other secondary outcomes)

Participants will be asked to:

* Complete a baseline assessment
* then use the self-help app for 5 weeks
* Complete a second assessment and participate in a short semi-structured interview regarding acceptability and feasibility.

Researchers will compare an intervention group to a wait-list control group to see if the use of the self-help app has an effect on secondary outcomes.

DETAILED DESCRIPTION:
This study examines the acceptance and feasibility of an app designed to provide self-help information to grieving Syrian refugees in Switzerland. The app solely offers information and tips for self-help for grieving individuals. Its goal is not to provide psychological treatment and does not replace psychological assistance from a professional.

The app was developed in close collaboration with the Swiss Red Cross (SRC), potential users, and experts to tailor it to the needs of grieving Syrian refugees. The app is designed to serve as a supplementary module for the SRC's Sui app after the completion of this study.

Developed in the Arabic language, the app consists of five chapters, each with several subchapters. These chapters cover various information on grief and grief reactions, tips, audio exercises, case vignettes, explanatory videos, video testimonials, as well as written information on various topics such as resources, the importance of social relationships, and daily structure.

Apart from the ability to read, understand, and write in Arabic, familiarity with using a smartphone, and access to the internet, no special skills or conditions are required for using the app.

The self-help program is available as an app on common iOS and Android devices. The app does not include invasive components or medications. It only provides information and general recommendations for grieving individuals. Users can input data into the app, but the app merely stores this information. The app does not manipulate data with the entered information (e.g., it does not provide personalized recommendations or feedback based on user inputs).

In this study, we aim to determine the feasibility and acceptability of this app for grieving Syrian refugees. Additionally, we want to assess whether there are fewer grief symptoms after using the app. The results of the app will help us further tailor it to the needs of the users. To investigate this, we are recruiting 30 study participants who will be randomly assigned to one of two groups. One group will use the app for 5 weeks, while the other group will wait for 5 weeks before gaining access to the app. Both groups will complete questionnaires at two measurement points, with the first group also being asked to provide feedback on the app in a brief interview.

ELIGIBILITY:
Inclusion Criteria:

* Syrian refugees living in Switzerland
* Min. 18 years old
* Able to give informed consent as documented by signature
* Can read and understand, as well as write Arabic
* Possess a smartphone with access to the internet
* Have experienced the loss of a loved one due to death at least 3 months ago
* Severity score of at least 3 in at least one item of the IPGDS

Exclusion Criteria:

* Acute suicidality measured by self-report
* Lack of knowledge of Arabic language, both spoken and/or written

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Intervention satisfaction | 5 weeks after baseline
  Client Satisfaction Questionnaire for Internet Interventions (CSQ-I). Items are rated from 1 to 4 (1= No' definitely not' 2= No' I don't think so' 3= Yes' I think so' 4=Yes' definitely), with higher scores indicating higher satisfaction.
Evaluation of the process | 5 weeks after baseline
  A short semi-structured interview was developed to assess the overall experience of the participants, the content of the intervention, the adherence to the intervention and the burden of the assessments.
Adherence | 5 weeks after baseline
  Number of modules that a person has completed

SECONDARY OUTCOMES:
Grief severity | Baseline and 5 weeks after baseline
  International ICD-11 Prolonged Grief Disorder Scale (IPGDS). Employs a 5-point scale: 1 = almost never (less than once a month), 2 = rarely (monthly), 3 = sometimes (weekly), 4 = often (daily), and 5 = always (several times a day), higher scores mean higher grief severity.
Depression | Baseline and 5 weeks after baseline
  Patient Health Questionnaire-9 Item (PHQ-9). Employs a scale ranging from 0 = never to 4 = practically every day. A higher score on the PHQ9 (range = 1 - 27) means a greater severity of depressive symptoms.
PTSD symptoms | Baseline and 5 weeks after baseline
  PTSD Checklist 5 8- item Version (PCL-5). Responses are scored on a scale from 0 to 4 with higher scores indicating more pronounced symptom severity.
Anxiety | Baseline and 5 weeks after baseline
  Generalized Anxiety Disorder Screener (GAD-7). Employs a scale ranging from 0 = never to 4 = practically every day. A higher score on the GAD-7 (range = 0 - 21) means a greater severity of anxiety symptoms.
Health and disability levels | Baseline and 5 weeks after baseline
  WHO Disability Assessment Scale 2.0 (WHODAS 2.0). Items are answered on a 5-point scale ranging from 0 = "none" to 4 = "extreme or cannot do".
Psychological well being | Baseline and 5 weeks after baseline
  WHO-5 Wellbeing Index (WHO-5). Items (e..g. "I have felt cheerful and in good spirits") are rated from 0="at no time" to 5="all the time".

OTHER OUTCOMES:
Life stressors of refugees | Baseline and 5 weeks after baseline
  Post Migration Living Difficulties Scale (PMLD; adapted to Swiss context). Items are rated on a five-point scale (0 not a problem to 4 very serious problem)
Perceived social support | Baseline and 5 weeks after baseline
  Multidimensional Scale of Perceived Social Support (MSPSS). Items are rated on a seven point scale (1 very strongly disagree to 7 very strongly agree), higher scores indicate higher perceived social support.
Voluntary qualitative feedback to individual chapters | 5 weeks after baseline
  Participants will have the possibility to input feedback concerning the content of individual chapters of the app during the app usage phase. This will be done through the app by including an open question after each chapter ("What feedback would you like to give us concerning the content of this previous chapter?")
Socio-demographic information | Baseline
  Sex, age, ethnicity, marital status, level of education, work situation, immigration status and time lived in Switzerland, loss-related characteristics such as the time of loss(es), the relationship to the deceased, the age and gender of lost person, cause of death, sudden or expected bereavement, ambiguous loss, information on whether currently undergoing psychotherapeutic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Thoma, PD Dr., Study Chair — University of Zurich; Anaïs Aeschlimann, MSc, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bech P, Olsen LR, Kjoller M, Rasmussen NK. Measuring well-being rather than the absence of distress symptoms: a comparison of the SF-36 Mental Health subscale and the WHO-Five Well-Being Scale. Int J Methods Psychiatr Res. 2003;12(2):85-91. doi: 10.1002/mpr.145. PMID 12830302
- [Background] Boss L, Lehr D, Reis D, Vis C, Riper H, Berking M, Ebert DD. Reliability and Validity of Assessing User Satisfaction With Web-Based Health Interventions. J Med Internet Res. 2016 Aug 31;18(8):e234. doi: 10.2196/jmir.5952. PMID 27582341
- [Background] Killikelly C, Zhou N, Merzhvynska M, Stelzer EM, Dotschung T, Rohner S, Sun LH, Maercker A. Development of the international prolonged grief disorder scale for the ICD-11: Measurement of core symptoms and culture items adapted for chinese and german-speaking samples. J Affect Disord. 2020 Dec 1;277:568-576. doi: 10.1016/j.jad.2020.08.057. Epub 2020 Aug 27. PMID 32896722
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lowe B, Kroenke K, Herzog W, Grafe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord. 2004 Jul;81(1):61-6. doi: 10.1016/S0165-0327(03)00198-8. PMID 15183601
- [Background] Price M, Szafranski DD, van Stolk-Cooke K, Gros DF. Investigation of abbreviated 4 and 8 item versions of the PTSD Checklist 5. Psychiatry Res. 2016 May 30;239:124-30. doi: 10.1016/j.psychres.2016.03.014. Epub 2016 Mar 8. PMID 27137973
- [Background] Schick M, Zumwald A, Knopfli B, Nickerson A, Bryant RA, Schnyder U, Muller J, Morina N. Challenging future, challenging past: the relationship of social integration and psychological impairment in traumatized refugees. Eur J Psychotraumatol. 2016 Feb 12;7:28057. doi: 10.3402/ejpt.v7.28057. eCollection 2016. PMID 26886484
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Üstün, T., Kostanjsek, N., Chatterji, S., & Rehm, J. (Hrsg.). (2010). Measuring health and disability: Manual for WHO Disability Assessment Schedule WHODAS 2.0. World Health Organization.
- [Background] Zimet, G., Dahlem, N., Zimet, S., & Farley, G. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52(1), 30-41. https://doi.org/10.1207/s15327752jpa5201_2